CLINICAL TRIAL: NCT05673889
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY TO EVALUATE THE EFFECT OF A SINGLE ORAL DOSE OF ARV-471 (PF-07850327) ON THE PHARMACOKINETICS OF DABIGATRAN IN HEALTHY PARTICIPANTS
Brief Title: A Study to Understand the Effect of a Study Medicine Called ARV-471 on Dabigatran Etexilate in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891008; 2022-003397-23 (EudraCT Number)
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabigatran etexilate with and without ARV-471 (Experimental): Dabigatran etexilate administered as a single dose in Period 1 and Period 2. ARV-471 administered as a single dose in Period 2.
  Interventions: Drug: ARV-471; Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: ARV-471 — Experimental
  Other Names: PF-07850327
Drug: Dabigatran etexilate — Probe substrate
  Other Names: PRADAXA®

SUMMARY:
The purpose of this study is to understand if ARV-471 affects how a medicine called, dabigatran etexilate, gets absorbed or processed into the body in healthy adults.

All participants in this study will receive one dose of dabigatran etexilate alone by mouth in Period 1. In Period 2, everyone will receive one dose of dabigatran etexilate by mouth approximately 90 minutes after receiving one dose of ARV-471 by mouth. The levels of dabigatran in Period 1 will be compared to the levels of dabigatran in Period 2. This will help us to determine if and how ARV-471 affects dabigatran gets absorbed into the body differently in healthy adults.

All participants will stay at the study clinic for approximately 8 days and 7 nights.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants of non-childbearing potential who are overtly healthy as determined by medical evaluation and are between the ages of 18 and 70 years, inclusive at the time of signing the informed consent document (ICD).
* Body mass index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Pregnant female participants, breastfeeding female participants, female participants of childbearing potential. Male participants with partners currently pregnant; male participants of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 90 days after the last dose of investigational product.
* Active bleeding or risk of bleeding including prior personal or familiar history of abnormal bleeding, hereditary or acquired coagulation or platelet disorder or abnormal coagulation test (PT/INR or PTT/aPTT greater than upper limit of normal) result at screening. Any significant risk factor for major bleeding and this may include but not limited to current or recent GI ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, or other conditions or situations related to COVID-19 pandemic that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription medications, including vitamins, dietary and herbal supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention or a longer washout is required for those that fall into the categories below:

  * Moderate or strong cytochrome P450 (CYP) 3A / P-glycoprotein (P-gp) inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
  * Moderate or strong CYP3A/P-gp inhibitors which are prohibited within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Standard 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 Periods in a single fixed sequence. Twenty-four participants were screened and passed. All 24 participants were assigned to the study treatment and all completed the study.
Groups:
- All Participants: Participants received a single oral dose of dabigatran etexilate (as mesylate) 75 milligram (mg) on Period 1 Day 1. A minimum washout period of 4 days was required after dabigatran etexilate (as mesylate) administration in Period 1. After completion of Period 1, participants received a single oral dose of ARV-471 (PF-07850327) 200 mg followed by a single oral dose of dabigatran etexilate (as mesylate) 75 mg on Period 2 Day 1.
Period: Period 1 (4 Days)
Arm/Group | All Participants
Started | 24
Completed | 24
Not Completed | 0
Period: Period 2 (3 Days)
Arm/Group | All Participants
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was defined as all participants enrolled and who took at least 1 dose of study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  Black or African American | 4
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Dabigatran When Dabigatran Etexilate is Administered Alone Versus When Dabigatran Etexilate is Administered With ARV-471
Description: Cmax was defined as maximum observed plasma concentration. Cmax for total dabigatran was observed directly from data.
Time Frame: Period 1 and 2: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose on Day 1
Population: Analysis population included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of primary interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Period 1: Dabigatran 75 mg: Participants received dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) on Period 1 Day 1.
- Period 2: Dabigatran 75 mg + ARV-471 200 mg: Participants received ARV-471 (as 2 tablets of 100 mg) and dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) on Period 2 Day 1.
Arm/Group | Period 1: Dabigatran 75 mg | Period 2: Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 24 | 24
nanogram per milliliter (ng/mL) | 49.80 (94) | 95.72 (66)
Statistical Analysis 1: Comparison: Period 1: Dabigatran 75 mg vs Period 2: Dabigatran 75 mg + ARV-471 200 mg; Dabigatran etexilate administered alone as Reference, ARV-471 coadministered with dabigatran etexilate as Test. Natural log transformed Cmax was analyzed using a mixed effect model with treatment as fixed effects and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 192.20, 90% CI 2-sided [166.56 to 221.79] — The ratios (and 90% CIs) are expressed as percentages

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Total Dabigatran When Dabigatran Etexilate is Administered Alone vs Dabigatran Etexilate is Administered With ARV-471
Description: AUCinf was defined as area under the concentration-time curve from time 0 extrapolated to infinity. AUCinf was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve; AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: Period 1 and 2: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Period 1: Dabigatran 75 mg | Period 2: Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 23 | 24
nanogram*hour per milliliter (ng*hr/mL) | 522.3 (42) | 949.6 (63)
Statistical Analysis 1: Comparison: Period 1: Dabigatran 75 mg vs Period 2: Dabigatran 75 mg + ARV-471 200 mg; [analysis description as in outcome 1, analysis 1]; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 197.81, 90% CI 2-sided [177.32 to 220.66] — The ratios (and 90% CIs) are expressed as percentages

3. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship with the study intervention. SAE is defined as one of the following: is fatal or life threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 5) of study intervention (up to 40 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Dabigatran 75 mg: Participants received dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) on Period 1 Day 1.
- Dabigatran 75 mg + ARV-471 200 mg: Participants received ARV-471 (as 2 tablets of 100 mg) and dabigatran etexilate (as mesylate) (as 1 capsule of 75 mg) on Period 2 Day 1.
Arm/Group | Dabigatran 75 mg | Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 24 | 24
Participants
  Participants with all-causality TEAEs | 6 | 6
  Participants with all-causality SAEs | 0 | 0
  Participants with treatment related TEAEs | 3 | 1
  Participants with treatment related SAEs | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid, cystatinC); electrolytes (sodium, potassium, chloride, calcium, bicarbonate); clinical chemistry (glucose); urinalysis (dipstick [decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, bilirubin], microscopy. Abnormality was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day -1) up to Period 2 Day 3 (8 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention and with at least 1 observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 75 mg | Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 24 | 24
Participants
  Monocytes/Leukocytes (%) >1.2 × ULN | 2 | 2
  Leukocyte Esterase >=1 | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs (blood pressure and pulse rate) were obtained with participant following at least a 5-minute rest in a supine position. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 3 (7 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 75 mg | Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 24 | 24
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria include a) a postdose QTc corrected using Fridericia's formula (QTcF) increased by >60 millisecond (ms) from the baseline and the absolute QTcF value >450 ms; or b) an absolute QTcF value >500 ms for any scheduled ECG.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 3 (7 days)
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 75 mg | Dabigatran 75 mg + ARV-471 200 mg
Number analyzed (Participants) | 24 | 24
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: From the first dose (Day 1) up to 35 days after the last dose (Day 5) of study intervention (up to 40 days).
Arm/Group | Period 1: Dabigatran 75 mg | Period 2: Dabigatran 75 mg + ARV-471 200 mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Dabigatran 75 mg (N=24) | Period 2: Dabigatran 75 mg + ARV-471 200 mg (N=24)
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Haematoma (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT05673889/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT05673889/SAP_001.pdf